CLINICAL TRIAL: NCT04721249
Title: A Randomized add-on Trial of D-serine for Depression
Brief Title: D-serine Supplementation for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: André Schmidt (Other)
Responsible Party: Sponsor-Investigator, André Schmidt, Principal Investigator, Psychiatric Hospital of the University of Basel
Organization: Psychiatric Hospital of the University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS-2124
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Active Comparator)
  Interventions: Dietary Supplement: D-serine
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: D-serine — Patients will receive four 500mg capsules of D-serine each day over a course of six weeks (two after breakfast and two after dinner).
  Arms: Verum
Dietary Supplement: Placebo — Patients in the placebo group will receive four placebo capsules each day (two after breakfast and two after dinner). The placebo capsules will contain Mannotol / Mannitol-Silica (99.5/0.5, respectively) and will be indistinguishable from D-serine by matching colour, shape, size and packaging.
  Arms: Placebo

SUMMARY:
The glutamate system is emerging as target for the development of novel antidepressant medication, in particular compounds modulating the NMDA receptor. While the NMDA receptor antagonist ketamine is an effective option for many treatment-restistant patients, it is also accompanied by dissociative and cognitive effects and also bears the risk to develop addiction, side effects that are significantly restricting its clinical utility. There is now compelling evidence of the antidepressant potential of D-serine, a NMDAR co-agonist. Compared to ketamine, D-serine goes along without any psychotomimetic effects or other side effects and thus might be a prom-ising novel antidepressant.

This study represents the first randomized control trial to test the efficacy of D-serine as an adjuvant therapy in patients with depression and thereby adds to re-cent efforts to establish novel glutamatergic antidepressants. Besides clinical measures, this study also explores the biological mechanisms underlying D-serine's clinical effect.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Inpatients with a diagnosis of MDD with a current moderate-to-severe episode (HAM-D score > 16) (7)
* Treatment as usual (TAU) for depression. TAU for depression may include no treatment at all or standard pharmacotherapy (antidepressants and antipsychotics such as aripiprazole, risperidone or quetiapine) and / or psychotherapy.
* Able to read and understand study procedures and participant's information

Exclusion Criteria:

* Other primary psychiatric diagnoses than MDD such as substance use and psychotic disorders
* Serious suicide attempts
* Contradiction for MRI (no pacemaker, MRI incompatible metal implants or splinters in the body, past heart/head surgery, past stroke/brain injury, claustrophobia)
* Pregnant or lactating women (pregnancy test)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Depression Severity | Change from baseline HAM-D score at 6 weeks
  measured with the Hamilton Depression Rating Scale (HAM-D)

SECONDARY OUTCOMES:
Anxiety | Change from baseline STAI score at 6 weeks
  measured with the State-and Trait-Anxiety Inventory (STAI)
Anhedonia | Change from baseline SHAPS score at 6 weeks
  measured with the Snaith-Hamilton-Pleasure Scale (SHAPS)
Neurocognition | Change from baseline VLMT score at 6 weeks
  measured with the Verbal Learning and Memory Test (VLMT)
Prefrontal glutamate concentration | Change from baseline glutamate level at 6 weeks
  measured with magnetic resonance spectroscopy (MRS)
Stress level | Change from baseline cortisol level at 6 weeks
  measured with Cortisol awakening responses
Inflammation | Change from baseline interleukin 1 and 6 level at 6 weeks
  measured with the blood levels of interleukin 1 and 6

CONTACTS AND LOCATIONS:
Overall Officials: André Schmidt, PD Dr, Principal Investigator — University of Basel, Department of Psychiatry (UPK)
Locations (1):
- University of Basel, Department of Psychiatry (UPK), Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sempach L, Schaub AC, Bruhl AB, Sterzer P, Lang UE, Schmidt A. Adjunctive d-serine treatment for major depressive disorder: A randomized clinical trial. J Affect Disord. 2025 Oct 15;387:119504. doi: 10.1016/j.jad.2025.119504. Epub 2025 May 26. PMID 40436209